CLINICAL TRIAL: NCT00210353
Title: Multicenter Randomized Trial of Chlorambucil Versus Chlorambucil Plus Rituximab Versus Rituximab in Extranodal Marginal Zone B-cell Lymphoma of Mucosa Associated Lymphoid Tissue (MALT Lymphoma)
Brief Title: Randomized Trial of Chlorambucil Versus Chlorambucil Plus Rituximab Versus Rituximab in MALT Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG19
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma, Mucosa-Associated Lymphoid Tissue
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Chlorambucil; Pharmaceutical Preparations; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM A (Active Comparator): chlorambucil 6 mg/m2 daily during the first 6 weeks of treatment; two weeks rest; chlorambucil 6 mg/m2 daily during the first two of a four weeks cycles (total of 4 cycles)
  Interventions: Drug: chlorambucil (drug)
- ARM B (Experimental): rituximab 375 mg/m2 iv, d1, d8, d15, d22 chlorambucil 6 mg/m2 os, daily during the first 6 weeks of treatment two weeks rest chlorambucil 6 mg/m2 os daily during the first two of a four weeks cycles (total of 4 cycles) rituximab 375 mg/m2 iv at day 1 of each cycle
  Interventions: Drug: rituximab+chlorambucil
- ARM C (Since April 2006) (Experimental): rituximab 375 mg/m2 iv on days 1, 8, 15, 22, 56, 84, 112, 140
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: chlorambucil (drug) — chlorambucil 6 mg/m2 daily during the first 6 weeks of treatment, two weeks rest, chlorambucil 6 mg/m2 daily during the first two of a four weeks cycles (total of 4 cycles)
  Arms: ARM A
Drug: rituximab+chlorambucil — rituximab 375 mg/m2 iv, d1, 8, 15, 22, chlorambucil 6 mg/m2 os, daily during the first 6 weeks of treatment, ; two weeks rest; chlorambucil 6 mg/m2 os, daily during the first two of a four weeks cycles (total of 4 cycles) rituximab 375 mg/m2 iv at day 1 of each cycle
  Arms: ARM B
Drug: rituximab — rituximab 375 mg/m2 iv on days 1, 8, 15, 22, 56, 84, 112, 140
  Arms: ARM C (Since April 2006)

SUMMARY:
Assess the therapeutic activity and safety of the combination of Chlorambucil and Rituximab in MALT lymphomas and determine whether the addition of Rituximab to Chlorambucil will improve the outcome of MALT lymphoma in comparison to treatment with Chlorambucil alone.

In April 2006, a third arm of treatment was added to compare the antitumor activity and safety of rituximab alone vs chlorambucil alone

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven diagnosis of CD20-positive marginal zone B-cell lymphoma of MALT type arisen at any extranodal site
2. any stage (Ann Arbor I-IV)
3. either de novo, or relapsed disease following local therapy (including surgery, radiotherapy and antibiotics for H. pylori-positive gastric lymphoma)
4. no evidence of histologic transformation to a high grade lymphoma
5. measurable or evaluable disease
6. age > 18
7. life expectancy of at least 1 year
8. ECOG performance status 0-2
9. no prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer
10. no prior chemotherapy
11. no prior immunotherapy with any anti-CD20 monoclonal antibody
12. no prior radiotherapy in the last 6 weeks
13. no corticosteroids during the last 28 days, unless prednisone chronically administered at a dose <20 mg/day for indications other than lymphoma or lymphoma-related symptoms
14. no evidence of clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months before study entry
15. no evidence of symptomatic central nervous system (CNS) disease
16. no impairment of bone marrow function (WBC >3.0x109/L, ANC >1.5x109/L, PLT >100x109/L), unless due to lymphoma involvement
17. no major impairment of renal function (serum creatinine <1,5x upper normal) or liver function (ASAT/ALAT <2,5 upper normal, total bilirubin <2,5x upper normal), unless due to lymphoma involvement
18. no evidence of active opportunistic infections
19. no known HIV infection
20. no active HBV and/or HCV infection
21. no pregnant or lactating status
22. appropriate contraceptive method in women of childbearing potential or men
23. absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
24. informed consent must be given according to national/local regulations before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2003-01; Primary Completion 2015-04 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, MD, Study Chair — International Extranodal Lymphoma Study Group/Oncology Institute of Southern Switzerland. Bellinzona; Emilio Montserrat, MD, Study Chair — Clinic Hospital Universitari, Hematology. Barcelona; Catherine Thieblemont, MD, Study Chair — Centre Hospitalier Lyon Sud, Hematology. Lyon; Giovanni Martinelli, MD, Study Chair — Hemato-oncology. European Oncology Institute. Milan; Peter Johnson, MD, Study Chair — Oncology Unit. Southampton General Hospital. Southampton; Maurizio Martelli, MD, Study Chair — Hematology. Università La Sapienza. Roma
Locations (75):
- Belgium (7):
  - ACZA Campus Stuivenberg, Antwerp
  - AZ StJan, Bruges
  - St Luc, Brussels
  - ULB Hopital Erasme, Brussels
  - CHNDRF, Charleroi
  - Hospital St Joseph, Gilly
  - UCL de Mont Godinne, Yvoir
- France (16):
  - Centre Hospitalier de Blois, Blois
  - Hopital Avicenne, Bobigny
  - CHU, Dijon
  - Centre Hospitalier, Lens
  - CHRU Lille, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Arnold Villeneuve, Monpellier
  - CHU, Nancy
  - CHU Hotel Dieu, Nantes
  - Centre R. Gauducheau, Nantes-St. Herblain
  - Hopital Henri-Mondor, Paris
  - Hopital St Louis, Paris
  - Necker, Paris
  - Centre Henri Becquerel, Rouen
- Italy (20):
  - Spedali Civili, Brescia
  - Azienda ULSS 15 Alta Padovana, Cittadella
  - IST, Genova
  - Humanitas, Milan
  - San Raffaele Hospital, Milan
  - IEO, Milan
  - INT, Milan
  - Policlinico, Modena
  - Ospedale Civile, Piacenza
  - A.O. Bianchi-Melacrino-Morelli, Divisione di Ematologia, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - S. Eugenio, Rome
  - Università Cattolica Sacro Cuore, Rome
  - Università La Sapienza, Rome
  - Sassuolo GISL, Sassuolo
  - AOU Senese, Siena
  - A.O.U. San Giovanni Battista-Molinette, S.C. Ematologia 2, Torino
  - Trani GISL, Trani
  - Ospedale di Circolo Fondazione Macchi, Varese
  - Policlinico GB Rossi, Verona
- Spain (5):
  - Clinic Hospital Universitari, Barcelona
  - Hopital Mataro', Barcelona
  - Hopital Santa Creu i Sant Pau, Barcelona
  - University Hospital, Salamanca
  - Joan XXIII, Tarragona
- IOSI, Bellinzona, Switzerland
- United Kingdom (26):
  - Aberdeen Royal Infirmary, Aberdeen
  - Heartlands, Birmingham
  - Victoria Hospital, Blackpool
  - Royal Cornwall Hospital, Cornwall
  - Darent Valley Hospital, Dartford
  - Royal Devon &Exeter Healtcare NHS Trust, Devon
  - Russels Hall Hospital, Dudley
  - Western General Hospital, Edinburgh
  - Medway Hospital, Gillingham
  - Raigmore Hospital, Inverness
  - Liverpool Royal Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - Barts & the London NHS Trust, London
  - Royal Marsden NHS Foundation Trust, London
  - St Georges, London
  - Christie Hospital, Manchester
  - Mount Vernon Hospital, Middlesex
  - James Paget Hospital, Norfolk
  - Queen Elisabeth, Norfolk
  - Nottingham City Hospital, Nottingham
  - John Radcliffe, Oxford
  - Conquest Hospital, Saint Leonard on Sea
  - Weston Park, Sheffield
  - Southampton General Hospital, Southampton
  - Sandwell General Hospital, West Bromwich
  - Worchestershire Acute Hospital NHS Trust, Worcester

REFERENCES:
- [Derived] Bommier C, Zucca E, Chevret S, Conconi A, Nowakowski G, Maurer MJ, Cerhan JR, Thieblemont C, Lambert J. Early complete response as a validated surrogate marker in extranodal marginal zone lymphoma systemic therapy. Blood. 2024 Feb 1;143(5):422-428. doi: 10.1182/blood.2023020984. PMID 37801707
- [Derived] Zucca E, Conconi A, Laszlo D, Lopez-Guillermo A, Bouabdallah R, Coiffier B, Sebban C, Jardin F, Vitolo U, Morschhauser F, Pileri SA, Copie-Bergman C, Campo E, Jack A, Floriani I, Johnson P, Martelli M, Cavalli F, Martinelli G, Thieblemont C. Addition of rituximab to chlorambucil produces superior event-free survival in the treatment of patients with extranodal marginal-zone B-cell lymphoma: 5-year analysis of the IELSG-19 Randomized Study. J Clin Oncol. 2013 Feb 10;31(5):565-72. doi: 10.1200/JCO.2011.40.6272. Epub 2013 Jan 7. PMID 23295789
- See also: Click here for more information about this study — http://www.ielsg.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 10 January 2003 to 07 July 2010
Groups:
- ARM A - Chlorambucil: Chlorambucil 6 mg/m2 daily during the first 6 weeks of treatment; two weeks rest; chlorambucil 6 mg/m2 daily during the first two of a four weeks cycles (total of 4 cycles)
- ARM B - Rituximab + Chlorambucil: rituximab 375 mg/m2 iv, d1, d8, d15, d22 chlorambucil 6 mg/m2 os, daily during the first 6 weeks of treatment two weeks rest chlorambucil 6 mg/m2 os daily during the first two of a four weeks cycles (total of 4 cycles) rituximab 375 mg/m2 iv at day 1 of each cycle
- ARM C (Since April 2006) - Rituximab: Rituximab 375 mg/m2 iv on days 1, 8, 15, 22, 56, 84, 112, 140
Period: Overall Study
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Rituximab
Started | 151 | 152 | 151
Completed | 113 | 107 | 125
Not Completed | 38 | 45 | 26

BASELINE CHARACTERISTICS:
Population: Evaluable patients
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Rituximab | Total
Number analyzed (Participants) | 131 | 132 | 138 | 401
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 80] | 59.5 [26 to 79] | 62.5 [27 to 81] | 61 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 68 | 74 | 204
  Male | 69 | 64 | 64 | 197
Region of Enrollment [Number; unit: participants]
  Belgium | 8 | 5 | 15 | 28
  Italy | 54 | 52 | 58 | 164
  United Kingdom | 18 | 23 | 19 | 60
  France | 39 | 40 | 41 | 120
  Switzerland | 3 | 3 | 5 | 11
  Spain | 9 | 9 | 0 | 18
Ann Arbor stage [Count of Participants; unit: Participants] — Stage I: Involvement of 1 LN region or localized involvement of a 1 extra-lymphatic organ/site Stage II: Involvement of 2 or more LN regions on the same side of the diaphragm or localized of 1 associated extra-lymphatic organ/site and its regional nodes Stage III: Involvement of LN regions on both sides of the diaphragm accompanied by localized involvement of an extra-lymphatic organ/site, by involvement of spleen or both.
  Stage IV: Disseminated involvement of 1 or more extra-lymphatic organs
  Participants
    Ann Arbor Stage > 2 | 53 | 59 | 63 | 175
    Ann arbor stage ≤ 2 | 78 | 73 | 75 | 226
B-symptoms [Count of Participants; unit: Participants] — B-symptoms refer to systemic symptoms of fever, night sweats, and weight loss which can be associated with both Hodgkin's lymphoma and non-Hodgkin's lymphoma
  Participants
    Presence of B-symptoms | 6 | 20 | 16 | 42
    Absence of B symptoms | 125 | 112 | 122 | 359
International Prognostic Index (IPI) risk [Count of Participants; unit: Participants] — Model for predicting outcomes in patients with aggressive non-Hodgkin's lymphoma on the basis of the patients' clinical characteristics before treatment.
  Prognostic factors are:
  Age (< 60 years vs. > 60 years) Serum LDH level (< normal vs > normal) Performance status (0,1 vs. 2-4) Tumor stage (I/II vs. III/IV) Extranodal involvement (< 1 site vs. > 1 site)
  Risk Groups are:
  Risk Factors 0 + 1 - IPI Low; Risk Factors 2 - IPI Low Intermediate; Risk Factors 3 - IPI High Intermediate; Risk Factors 4 + 5 - IPI High.
  Participants
    Low | 79 | 74 | 76 | 229
    Low-intermediate | 25 | 34 | 35 | 94
    Intermediate-high | 23 | 20 | 25 | 68
    High | 3 | 4 | 2 | 9
    NA | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free-survival (EFS)
Description: Percentage of patients without events (failure of treatment or Death from any cause) after 5 years from trial registration
Time Frame: 5 years
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Rituximab
Number analyzed (Participants) | 131 | 132 | 138
percentage of patients | 51 [42 to 60] | 68 [60 to 76] | 51 [42 to 60]

2. Secondary Outcome: Complete and Partial Remission Rate - Percentage of Patients With Complete and Partial Response at the End of Treatment
Description: Response criteria were defined according to the NCI standardized response criteria for non-Hodgkin's lymphoma.
  Complete response. Disappearance of all detectable clinical and radiographic evidence of disease, disappearance of all disease-related symptoms, if present before therapy, and normalization of those biochemical abnormalities definitely assignable to NHL. Regression of all lymph nodes and nodal masses to normal (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm before therapy and to ≤ 1 cm for nodes that were 1.1-1.5 cm. Regression by more than 75% in the sum of the products of the greatest diameters).
  Partial response. Decrease by at least 50% in SPD of the six largest measurable lesions. It is not necessary for all lesions to have regressed to qualify for partial response, but no lesion should have progressed and no new lesion should appear.
  For primary gastric sites, response was based on GELA histologic grading system.
Time Frame: End of treatment (after 24 weeks of therapy)
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Rituximab
Number analyzed (Participants) | 131 | 132 | 138
percentage of patients | 85.5 [78.3 to 91.0] | 94.7 [89.4 to 97.8] | 78.3 [70.4 to 84.8]

3. Secondary Outcome: Response Duration (Time to Relapse or Progression) - Percentage of Patients in Continuous Remission at Five Years From Trial Registration
Description: Response criteria were defined according to the NCI standardized response criteria for non-Hodgkin's lymphoma.
  Complete response (CR). Disappearance of all detectable clinical and radiographic evidence of disease, disappearance of all disease-related symptoms, if present before therapy, and normalization of those biochemical abnormalities definitely assignable to NHL. Regression of all lymph nodes and nodal masses to normal (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm before therapy and to ≤ 1 cm for nodes that were 1.1-1.5 cm. Regression by more than 75% in the sum of the products of the greatest diameters).
Time Frame: 5 years
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Rituximab
Number analyzed (Participants) | 131 | 132 | 138
percentage of patients | 70 [60 to 78] | 79 [71 to 85] | 66 [56 to 74]

4. Secondary Outcome: Progression-free-survival (PFS)
Description: Percentage of patients without disease progression after 5 years from trial registration
Time Frame: 5 years
Population: Evaluable Patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- ARM C (Since April 2006) - Ritiximab: rituximab 375 mg/m2 iv on days 1, 8, 15, 22, 56, 84, 112, 140
Arm/Group | ARM A - Chlorambucil | ARM B - Rituximab + Chlorambucil | ARM C (Since April 2006) - Ritiximab
Number analyzed (Participants) | 131 | 132 | 138
percentage of patients | 59 [50 to 68] | 72 [63 to 79] | 57 [48 to 65]

5. Secondary Outcome: Overall Survival
Description: Percentage of patients alive after 5 years from trial registration
Time Frame: 5 years
Population: Evaluable Patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ARM A | ARM B | ARM C (Since April 2006)
Number analyzed (Participants) | 131 | 132 | 138
percentage of patients | 89 [82 to 93] | 90 [83 to 94] | 92 [86 to 96]

ADVERSE EVENTS:
Time Frame: Seven years and eight months
Arm/Group | ARM A | ARM B | ARM C (Since April 2006)
All-Cause Mortality (participants affected / at risk) | 20/131 | 25/132 | 13/138
Serious Adverse Events (participants affected / at risk) | 4/131 | 20/132 | 13/138
Other Adverse Events (participants affected / at risk) | 42/131 | 77/132 | 59/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (N=131) | ARM B (N=132) | ARM C (Since April 2006) (N=138)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal Cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Injection site thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stent removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2)
metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic reactions (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease prpgression NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (N=131) | ARM B (N=132) | ARM C (Since April 2006) (N=138)
Fatigue (General disorders) | 16 (16) | 13 (13) | 16 (16)
Pyrexia (General disorders) | 1 (1) | 6 (6) | 9 (9)
Nausea (Gastrointestinal disorders) | 7 (7) | 18 (18) | 7 (7)
Infection (Infections and infestations) | 17 (17) | 13 (13) | 14 (14)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 11 (11) | 7 (7)
Infusion related reactions (General disorders) | 0 (0) | 21 (21) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No